CLINICAL TRIAL: NCT00222443
Title: Pilot Study Combining Temozolomide, Oncovin, Camptosar and Oral Antibiotic in Children and Adolescents With Recurrent Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JEC Toca One; NCT00277719 (obsolete NCT alias)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Lymphomas; Tumors
Keywords: Recurrent solid tumors; recurrent lymphomas; Pediatrics; Adolescents
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — Irinotecan

INTERVENTIONS:
Drug: Irinotecan

SUMMARY:
Determine toxicity and maximum tolerated dose of escalating daily protracted irinotecan, with weekly vincristine, temozolomide and vantin; to evaluate the feasibility of repetitive cycles of this chemotherapy and to estimate the response rate to this combination in children and adolescents with recurrent solid tumors and lymphomas.

DETAILED DESCRIPTION:
Determine toxicity and maximum tolerated dose of escalating daily protracted irinotecan, with weekly vincristine, temozolomide and vantin; to evaluate the feasibility of repetitive cycles of this chemotherapy and to estimate the response rate to this combination in children and adolescents with recurrent solid tumors and lymphomas.

Temozolomide is given by mouth one hour prior to each daily irinotecan dose days 1-5 of each cycle. 100 mg/m2/day. Irinotecan is given IV in dose escalation (minimum of 3 and up to 6 patients per cohort) starting at 15 mg/m2/day daily for 5 days for 2 weeks. Vincristin is given IV 1.5 mg/m2/dose (max dose 2mg) days 1 and 8 of each cycle. Vantin is given 10 mg/kg/day divided in 2 oral doses (max dose 400 mg/day) started 48 hours prior to the start of each treatment cycle and continued for 48 hours after last irinotecan dose. Cycle repeated every 28 days.

Therapy will continue for a minimum of two cycles unless there is progression of disease or unacceptable toxicity and may be continued as long as patient tolerates therapy and there is continued disease control up to one year of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Under age 21 years at time of study entry
* Malignant solid tumor, including CNS tumors and lymphomas
* Recurrent or refractory disease not amenable to other potentially curative therapies
* At least three weeks since last myelosuppressive chemotherapy > 6 months from allogeneic stem cell transplant
* Adequate renal and hepatic function
* Adequate peripheral blood counts unless bone marrow is involved

Exclusion Criteria:

* Patients with leukemia not eligible
* Patients with uncontrolled infection excluded
* Patients who have received more than 4 prior chemotherapies
* Patients who are receiving P450 enzyme-inducing anticonvulsants
* Patients who are receiving any other cancer chemotherapy or any other investigational agent
* Possible pregnancy will be excluded

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Determine toxicity and maximum tolerated dose of escalating daily protracted irinotecan.
Evaluate feasibility of repetitive cycles of this combination .

SECONDARY OUTCOMES:
Estimate response rate in children and adolescents with recurrent solid tumors and lymphomas.

CONTACTS AND LOCATIONS:
Overall Officials: William H Meyer, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Oklahoma University Health Sciences Center-Jimmy Everest Center, Oklahoma City, Oklahoma, United States